CLINICAL TRIAL: NCT05107752
Title: Stellate Ganglion Block to Augment Trauma-focused Therapy Among Veterans With PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: The Stellate Institute (Unknown); Navy SEAL Foundation (Unknown)
Responsible Party: Principal Investigator, Craig Bryan, Stress, Trauma, and Resilience (STAR) Professor, Ohio State University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2021H0228
Record Dates: First submitted 2021-10-14; First posted 2021-11-04 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: PTSD; Trauma and Stressor Related Disorders; Trauma, Psychological; Post Traumatic Stress Disorder
Keywords: veteran; military; stellate ganglion block; cognitive processing therapy; cognitive behavioral therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Trauma and Stressor Related Disorders; Psychological Trauma

STUDY DESIGN:
Intervention Model Description: All participants receive cognitive processing therapy during weeks 1 and 2. Participants will be randomly allocated to receive SGB during or 3 months after CPT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Stellate ganglion block (SGB) treatment during cognitive processing therapy (CPT) (Experimental): Participants will receive 12 sessions of cognitive processing therapy (CPT) for PTSD combined with SGB during the first week of CPT.
  Interventions: Behavioral: Cognitive Processing Therapy (CPT); Drug: Stellate Ganglion Block
- SGB three months after completing CPT (Experimental): Participant will receive 12 sessions of cognitive processing therapy (CPT) for PTSD and will receive SGB three months after completing the CPT sessions.
  Interventions: Behavioral: Cognitive Processing Therapy (CPT); Drug: Stellate Ganglion Block

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy (CPT) — Cognitive processing therapy (CPT) is a specific type of cognitive behavioral therapy that has been effective in reducing symptoms of PTSD that have developed after experiencing a variety of traumatic events including child abuse, combat, rape and natural disasters. CPT is generally delivered over 12 sessions and helps patients learn how to challenge and modify unhelpful beliefs related to the trauma. In so doing, the patient creates a new understanding and conceptualization of the traumatic event so that it reduces its ongoing negative effects on current life. This treatment is strongly recommended for the treatment of PTSD.
Drug: Stellate Ganglion Block — SGB is a procedure that has demonstrated efficacy for the reduction of PTSD symptoms. SGB is performed using real-time ultrasonography with an in-plane technique, and consists of 7-10 mL of ropivacaine 0.5%, which is injected around and into the site of the ganglion at the level of the C4 and C6 anterior tubercle (Mulvaney, Curtis et al., 2020). Ropivacaine is a long-acting amide local anesthetic agent and a pure S-enantiomer with a high pKa and relatively low solubility. Patients are not sedated during the procedure. Successful sympathetic blockade is confirmed by the presence of Horner's syndrome, which is characterized by constriction of the pupil (miosis) and drooping of the upper eyelid (ptosis). If Horner's syndrome is not observed within 20 minutes of the first injection, the right-sided SGB is repeated one hour later using the same technique. If Horner's syndrome is not confirmed after the second injection, no additional injections are provided.

SUMMARY:
Our long-term goal is to improve clinical outcomes among patients receiving psychological treatment for posttraumatic stress disorder (PTSD). The primary objective of this project is to examine if stellate ganglion block (SGB) improves outcomes among military personnel and veterans receiving cognitive processing therapy (CPT), an empirically-supported psychological treatment for PTSD. To accomplish this objective, we will enroll adult military personnel and veterans with a current diagnosis of PTSD and/or subthreshold PTSD, provide CPT sessions over two weeks, administer SGB during or after CPT, and repeatedly assess key outcomes during follow-up.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is the most frequently diagnosed mental health condition among veterans (Tanielian & Jaycox, 2008), with estimated rates of the condition ranging from 5-20% (Hoge, Castro, et al., 2004; Hoge, Terhakopian, et al., 2007; Milliken, Auchterlonie, & Hoge, 2007; Tanielian & Jaycox, 2008). PTSD is not just a consequence of combat, however; many military personnel and veterans experience noncombat-related traumas such as sexual assault and domestic abuse, or have histories of early life trauma such as child abuse that can also contribute to PTSD. Regardless of the associated event, PTSD is associated with a host of functional problems and negative outcomes among military personnel including occupational and marital dissatisfaction, violence, alcohol and substance abuse, and suicide (Hoge et al., 2004; Jakupcak et al., 2007; Panagioti, Gooding, & Tarrier, 2009).

Cognitive behavioral treatments are the most highly efficacious treatments for PTSD. Cognitive Processing Therapy (CPT) is one such treatment that has garnered a significant amount of empirical support, with a recent metaanalysis showing it was the most effective treatment for PTSD (Watts et al., 2013), typically yielding a 50% or larger reduction in PTSD symptoms from pre- to posttreatment. Despite CPT's effectiveness, a significant percentage of military veterans continue to experience moderate to severe symptoms afterwards, and nearly half continue to meet full criteria for the diagnosis (Harik, Grubbs, & Schnurr, 2016). Novel strategies for improving treatment outcomes are therefore needed.

Accumulating evidence supports the effectiveness of stellate ganglion block (SGB) for the treatment of PTSD. SGB is a procedure in which an injection of a long-acting local anesthetic, using ultrasound or fluoroscopic guidance, is made in the right side of the neck around the cervical sympathetic chain that controls the "fight or flight" response (the sympathetic nervous system). The cervical sympathetic chain is a two-way conduit that connects the parts of the brain that control the fight or flight response to the rest of the body. By blocking or "turning off" the cervical sympathetic chain, it is believed that the parts of the brain that control the fight or flight response are allowed to completely reset, resulting in long-term relief of the associated anxiety symptoms. Originally developed for the treatment of pain conditions, multiple case series have shown that right-sided SGB is associated with significant reductions in PTSD symptoms after SGB (Alino et al., 2013; Hickey et al., 2012; Lipov et al., 2008; Mulvaney et al., 2010, 2014), especially negative mood and hyperarousal symptoms (Lynch et al., 2016). Results of a recent randomized controlled trial in which SGB was compared to sham treatment further support the procedure's efficacy (Olmsted et al., 2019). In that study, PTSD symptom reduction in the SGB group was twice as large as the sham group. Research also supports SGB's safety and acceptability among patients with combat-related PTSD (McLean, 2015).

To date, however, the effectiveness of SGB when delivered in combination with first-line PTSD treatments like CPT has not been examined. The present study is designed to examine this issue from two perspectives. First, we will examine if the administration of SGB during CPT leads to larger reductions in PTSD symptoms as compared to CPT alone. Second, we will examine if the administration of SGB after CPT leads to significant reductions in PTSD symptoms among veterans who continue to experience moderate to severe symptoms after completing the therapy. To achieve this the study entails a single-blind, randomized clinical trial with wait list control. All participants will receive cognitive processing therapy (CPT), an empirically-supported psychological (non-medication) treatment for PTSD. Participants will be randomly assigned to receive stellate ganglion block (SGB) treatment at one of two time points: (1) during CPT or (2) three months after completing CPT. Outcomes will be assessed repeatedly for six months postbaseline.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Prior or current service in the U.S. military
* Diagnosis of PTSD within the last month
* Ability to speak and understand the English language
* Stable psychotropic medication dosing for at least 3 months
* Ability to complete the informed consent process

Exclusion Criteria:

* Prior SGB treatment or CPT treatment
* History of schizophrenia, another psychotic disorder, or bipolar disorder
* Moderate or severe traumatic brain injury
* Moderate or severe symptoms of a substance use disorder within the preceding 30 days
* Severe suicide risk warranting suicide-focused treatment and/or inpatient hospitalization
* Impaired mental status that precludes the ability to provide informed consent
* Any ongoing stressor or condition deemed by the investigators to place the participant at risk for injury or a poor outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptom severity | Screening, Week 0, Week 1, Week 2, Week 4, Week 8, Week 12, Week 13, Week 14, Week 16, Week 20, Week 24, Week 52
  PTSD symptom severity will be assessed using PTSD PCL-5. The scale includes 20 items that rate the severity of each symptom using a 5-point scale, with items summed to provide an overall metric of PTSD symptom severity.

SECONDARY OUTCOMES:
Change in depression symptom severity | Screening, Week 0, Week 1, Week 2, Week 4, Week 8, Week 12, Week 13, Week 14, Week 16, Week 20, Week 24, Week 52
  Severity will be measured using the Patient Health Questionnaire-9 (PHQ-9). The scale includes 9 items that rate the severity of each symptom using a 4-point scale, with items summed to provide an overall metric of depression symptom severity.
Change in anxiety symptom severity | Screening, Week 0, Week 1, Week 2, Week 4, Week 8, Week 12, Week 13, Week 14, Week 16, Week 20, Week 24, Week 52
  Severity will be measured using the Generalized Anxiety Disorder-7 (GAD-7) scale. The scale includes 7 items that rate the severity of each symptom using a 4-point scale, with items summed to provide an overall metric of anxiety symptom severity.
Change in somatic symptoms | Screening, Week 0, Week 1, Week 2, Week 4, Week 8, Week 12, Week 13, Week 14, Week 16, Week 20, Week 24, Week 52
  Symptoms will be measured using the Patient Health Questionnaire-15 (PHQ-15). The PHQ-15 is designed to assess the severity of 15 somatic/physical symptoms using a 3-point scale. Items can be summed to provide an overall metric of somatic symptoms and side effects.
Change in good end-state functioning | Screening, Week 0, Week 1, Week 2, Week 4, Week 8, Week 12, Week 13, Week 14, Week 16, Week 20, Week 24, Week 52
  Good end-state functioning is defined as having very low symptoms of both PTSD and depression, and is operationalized as a PCL-5 total score < 20 and a PHQ-9 total score < 10. It will be measured using a combination of these scores.

CONTACTS AND LOCATIONS:
Overall Officials: Craig J Bryan, PsyD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers interested in using IPD and/or computer code collected or generated as part of this study may do so by contacting the study PI. Researchers will be asked to complete a Data Use Request Form, which includes contact information, description of the research project for which the data and/or code would be used, specification of which data and/or code would be needed for their proposed project, an approximate time line for their proposed project, and authorship on their proposed project.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication of primary results
Access Criteria: All requests for data and/or code use will be reviewed by the PIs and co-Is and a majority vote will be used to determine whether the request is approved or not. If the request is approved, Dr. Bryan will inform the requestor, return a signed copy of the completed Data Use Request Form to the requestor, and let the requestor know that written IRB approval of the requestor's proposed study from the requestor's home institution will be required before data and/or code will be shared with the requestor. If a request is approved pending revision to the Data Use Request Form, Dr. Bryan will work with requestors to revise sections of their Data Use Request Forms in order to obtain approval. If the request is not approved, Dr. Bryan will inform the requestor and returned a signed copy of the completed Data Use Request Form to the requestor that includes an explanation for the denial.

REFERENCES:
- [Background] Alino J, Kosatka D, McLean B, Hirsch K. Efficacy of stellate ganglion block in the treatment of anxiety symptoms from combat-related post-traumatic stress disorder: a case series. Mil Med. 2013 Apr;178(4):e473-6. doi: 10.7205/MILMED-D-12-00386. PMID 23707834
- [Background] Harik, J. M., Grubbs, K. G., & Schnurr, P. P. (2016, November). Using graphics to communicate information about PTSD treatment effectiveness to patients. In J. L. Hamblen (Chair), Enhancing the quality of online information to support PTSD treatment engagement. Symposium presented at the 30th annual meeting of the International Society for Traumatic Stress Studies in Dallas, TX.
- [Background] Hicky A, Hanling S, Pevney E, Allen R, McLay RN. Stellate ganglion block for PTSD. Am J Psychiatry. 2012 Jul;169(7):760. doi: 10.1176/appi.ajp.2012.11111729. No abstract available. PMID 22760192
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems, and barriers to care. N Engl J Med. 2004 Jul 1;351(1):13-22. doi: 10.1056/NEJMoa040603. PMID 15229303
- [Background] Hoge CW, Terhakopian A, Castro CA, Messer SC, Engel CC. Association of posttraumatic stress disorder with somatic symptoms, health care visits, and absenteeism among Iraq war veterans. Am J Psychiatry. 2007 Jan;164(1):150-3. doi: 10.1176/ajp.2007.164.1.150. PMID 17202557
- [Background] Jakupcak M, Conybeare D, Phelps L, Hunt S, Holmes HA, Felker B, Klevens M, McFall ME. Anger, hostility, and aggression among Iraq and Afghanistan War veterans reporting PTSD and subthreshold PTSD. J Trauma Stress. 2007 Dec;20(6):945-54. doi: 10.1002/jts.20258. PMID 18157891
- [Background] Lipov EG, Joshi JR, Lipov S, Sanders SE, Siroko MK. Cervical sympathetic blockade in a patient with post-traumatic stress disorder: a case report. Ann Clin Psychiatry. 2008 Oct-Dec;20(4):227-8. doi: 10.1080/10401230802435518. No abstract available. PMID 19034755
- [Background] Lynch JH, Mulvaney SW, Kim EH, de Leeuw JB, Schroeder MJ, Kane SF. Effect of Stellate Ganglion Block on Specific Symptom Clusters for Treatment of Post-Traumatic Stress Disorder. Mil Med. 2016 Sep;181(9):1135-41. doi: 10.7205/MILMED-D-15-00518. PMID 27612365
- [Background] McLean B. Safety and Patient Acceptability of Stellate Ganglion Blockade as a Treatment Adjunct for Combat-Related Post-Traumatic Stress Disorder: A Quality Assurance Initiative. Cureus. 2015 Sep 10;7(9):e320. doi: 10.7759/cureus.320. PMID 26487996
- [Background] Milliken CS, Auchterlonie JL, Hoge CW. Longitudinal assessment of mental health problems among active and reserve component soldiers returning from the Iraq war. JAMA. 2007 Nov 14;298(18):2141-8. doi: 10.1001/jama.298.18.2141. PMID 18000197
- [Background] Mulvaney SW, Curtis KE, Ibrahim TS (2020) Comparison C6 Stellate Ganglion versus C6 and C4 Cervical Sympathetic Chain Blocks for Treatment of Posttraumatic Stress Disorder (PTSD): Analysis of 147 Patients. J Neurol Disord Stroke 7(3): 1163.
- [Background] Mulvaney SW, Lynch JH, Hickey MJ, Rahman-Rawlins T, Schroeder M, Kane S, Lipov E. Stellate ganglion block used to treat symptoms associated with combat-related post-traumatic stress disorder: a case series of 166 patients. Mil Med. 2014 Oct;179(10):1133-40. doi: 10.7205/MILMED-D-14-00151. PMID 25269132
- [Background] Mulvaney SW, McLean B, de Leeuw J. The use of stellate ganglion block in the treatment of panic/anxiety symptoms with combat-related post-traumatic stress disorder; preliminary results of long-term follow-up: a case series. Pain Pract. 2010 Jul-Aug;10(4):359-65. doi: 10.1111/j.1533-2500.2010.00373.x. Epub 2010 Apr 20. PMID 20412504
- [Background] Rae Olmsted KL, Bartoszek M, Mulvaney S, McLean B, Turabi A, Young R, Kim E, Vandermaas-Peeler R, Morgan JK, Constantinescu O, Kane S, Nguyen C, Hirsch S, Munoz B, Wallace D, Croxford J, Lynch JH, White R, Walters BB. Effect of Stellate Ganglion Block Treatment on Posttraumatic Stress Disorder Symptoms: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Feb 1;77(2):130-138. doi: 10.1001/jamapsychiatry.2019.3474. PMID 31693083
- [Background] Panagioti M, Gooding P, Tarrier N. Post-traumatic stress disorder and suicidal behavior: A narrative review. Clin Psychol Rev. 2009 Aug;29(6):471-82. doi: 10.1016/j.cpr.2009.05.001. Epub 2009 Jun 8. PMID 19539412
- [Background] Tanielian, T., & Jaycox, L.H. (2008). Invisible Wounds of War. Rand Corporation, 1-66.
- [Background] Watts BV, Schnurr PP, Mayo L, Young-Xu Y, Weeks WB, Friedman MJ. Meta-analysis of the efficacy of treatments for posttraumatic stress disorder. J Clin Psychiatry. 2013 Jun;74(6):e541-50. doi: 10.4088/JCP.12r08225. PMID 23842024